CLINICAL TRIAL: NCT01320696
Title: A Randomized, Double Blind, Multi-center, Phase 1/2 Study to Assess Safety and Immunogenicity of Five Dose Levels of a Reverse Genetic (RG) Reassortant H9N2 Pandemic Influenza Vaccine in Healthy Subjects Aged 18 to 49 Years
Brief Title: Reverse Genetic H9N2 Influenza Vaccine Study in Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 831001
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Results first posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): 50 subjects will be randomized 1:1:1:1:1 to 5 dose groups (10 subjects per treatment group) to receive 2 intramuscular injections of RG reassortant A/H9N2 influenza vaccine on Day 1 and Day 22
  Interventions: Biological: Reverse Genetic (RG) reassortant A/H9N2 influenza vaccine
- Cohort 2 (Experimental): After a safety data review of the first 50 subjects, a further 225 subjects will be randomized 1:1:1:1:1 to 5 dose groups and will receive 2 intramuscular injections of RG reassortant A/H9N2 influenza vaccine on Day 1 and Day 22
  Interventions: Biological: Reverse Genetic (RG) reassortant A/H9N2 influenza vaccine

INTERVENTIONS:
Biological: Reverse Genetic (RG) reassortant A/H9N2 influenza vaccine — Two intramuscular vaccinations; 5 dose groups: 3.75 µg, 7.5 µg, 15 µg, 30 µg or 45 µg HA antigen (strain A/H9N2/chicken/Hong Kong/G9/97; non-adjuvanted formulation

SUMMARY:
The purpose of the study is to identify the optimal dose level of a reverse genetic (RG) reassortant H9N2 pandemic influenza vaccine for further product development.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 to 49 years of age, inclusive, on the day of screening
* Subject has an understanding of the study and its procedures, agrees to its provisions, and gives written informed consent prior to study entry
* Subject is generally healthy, as determined by the investigator's clinical judgement through collection of medical history and performance of a physical examination
* Subject is physically and mentally capable of participating in the study as determined by the investigator
* Subject agrees to keep a daily record of symptoms for the duration of the study
* If female of childbearing potential, subject presents with a negative urine pregnancy test within 24 hours prior to first vaccination and agrees to employ adequate birth control measures for the duration of the study. For the purposes of this study at least one of the following types of US Food and Drug Administration (FDA) approved birth control measures shall be applied through completion of the Day 181 study visit:

  * Hormonal types of birth control (such as implants or birth control pills) or an intrauterine device
  * A barrier type of birth control measure (i.e. condoms, diaphragms, cervical caps, etc.)

Exclusion Criteria:

* Subject has a history of exposure to H9N2 influenza virus or a history of vaccination with an H9N2 influenza vaccine
* Subject is at potential occupational risk of contracting H9N2 influenza infection (e.g. poultry workers)
* Subject currently suffers from or has a history of a significant (requiring hospitalization or change in intervention in past 6 months)neurological, cardiovascular, pulmonary (including asthma), hepatic, rheumatic, autoimmune, hematological, metabolic or renal disorder such as but not limited to: multiple sclerosis, lupus, Guillain-Barre syndrome as determined by the investigator
* Subject has a body temperature of >= 100.4 degrees Fahrenheit (>= 38.0 degrees Celsius) on the day of vaccination, by oral measurement. [NOTE: Subjects meeting this exclusion criterion may be rescheduled for vaccination and study entry at a later date provided: 1) body temperature measured orally has decreased to < 100.4 degrees Fahrenheit (< 38.0 degrees Celsius); 2) all other inclusion/exclusion criteria are met; 3) the rescheduled date is no more than 14 days past the initial screening assessments and date; and 4) the study site is still enrolling subjects and randomization is not closed]
* Subject has a Body Mass Index (BMI) >= 35
* Subject has hypertension at screening that is graded as greater than Stage 1 (defined as a systolic pressure > 159 or diastolic pressure > 99 while seated and at rest (measurement shall be repeated twice before subject is excluded)
* Subject has clinically significant abnormal laboratory values at screening as determined by the investigator
* Subject tests positive for Human Immunodeficiency Virus (HIV), Hepatitis B surface Antigen (HBsAgs) or Hepatitis C Virus (HCV)
* Subject has any medically diagnosed or suspected immune deficient condition based on medical history and physical examination as determined by the investigator
* Subject has an immune compromising condition or disease, or is currently undergoing a form of treatment or was undergoing a form of treatment within 30 days prior to study entry that can be expected to influence immune response. Such treatment includes, but is not limited to, systemic or high dose inhaled (> 800 μg/day of beclomethasone dipropionate or equivalent) corticosteroids, radiation treatment or other immunosuppressive or cytotoxic drugs (use of inhaled and nasal steroids will be permitted)
* Subject has a history of severe (required immediate medical life threatening treatment and/or hospitalization) allergic reactions or anaphylaxis as determined by the investigator
* Subject has a rash, dermatologic condition or tattoos which may interfere with injection site reaction rating as determined by the investigator
* Subject has received any blood products (e.g. blood transfusion or immunoglobulins) within 90 days prior to study entry
* Subject has donated one or more units of blood (approximately 450 mL) or plasma within 30 days prior to study entry
* Subject has received any live vaccine within 4 weeks or an inactivated vaccine or a subunit vaccine within 2 weeks prior to vaccination in this study
* Subject has a functional or surgical asplenia
* Subject has a positive urine drug screen (unless the subject is currently prescribed the drug detected by a licensed health care provider and the continued administration of the drug would not otherwise exclude the subject from participation)
* Subject has a known or suspected problem with alcohol or drug abuse as determined by the investigator
* Subject is currently enrolled or has participated in another clinical study involving an investigational products (IP) or device within 30 days prior to study enrollment or is scheduled to participate in another clinical study involving an IP or device during the course of this study
* Subject is a member of the team conducting this study or is in a dependent relationship with one of the study team members. Dependent relationships include close relatives (i.e. children, partner/spouse, siblings, parents) as well as employees of the investigator or site personnel conducting the study
* If female, subject is pregnant or lactating at the time of study enrollment
* Any condition that in the opinion of the investigator would interfere with evaluation of the vaccine or interpretation of study results

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 353 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Izay, MD, Study Director — Baxter Innovations GmbH
Locations (5):
- United States (5):
  - Accelovance, Huntsville, Alabama
  - Accelovance, Melbourne, Florida
  - Accelovance, Peoria, Illinois
  - Accelovance, South Bend, Indiana
  - Accelovance, Rockville, Maryland

REFERENCES:
- [Derived] Aichinger G, Grohmann-Izay B, van der Velden MV, Fritsch S, Koska M, Portsmouth D, Hart MK, El-Amin W, Kistner O, Barrett PN. Phase I/II randomized double-blind study of the safety and immunogenicity of a nonadjuvanted vero cell culture-derived whole-virus H9N2 influenza vaccine in healthy adults. Clin Vaccine Immunol. 2015 Jan;22(1):46-55. doi: 10.1128/CVI.00275-14. Epub 2014 Oct 29. PMID 25355797

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 353 enrolled participants, 275 met inclusion criteria and were randomized to treatment.
Groups:
- 3.75 µg; 7.5 µg; 15 µg; 30 µg; 45 µg: Subjects to receive 2 intramuscular injections of Reverse Genetic (RG) reassortant A/H9N2 influenza vaccine on Day 1 and Day 22
Period: Overall Study
Arm/Group | 3.75 µg | 7.5 µg | 15 µg | 30 µg | 45 µg
Started | 56 | 55 | 54 | 55 | 55
Vaccinated Vacc. 1 | 56 | 55 | 54 | 55 | 55
Vaccinated Vacc. 2 | 53 | 53 | 54 | 55 | 54
Completed | 51 | 51 | 51 | 50 | 52
Not Completed | 5 | 4 | 3 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3.75 µg | 7.5 µg | 15 µg | 30 µg | 45 µg | Total
Number analyzed (Participants) | 56 | 55 | 54 | 55 | 55 | 275
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (8.6) | 32.6 (8.7) | 33.8 (8.1) | 35.8 (9.3) | 34.1 (9.0) | 33.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 27 | 31 | 31 | 29 | 151
  Male | 23 | 28 | 23 | 24 | 26 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 2 | 4 | 4 | 19
  Not Hispanic or Latino | 52 | 50 | 52 | 51 | 51 | 256
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 1 | 2 | 2 | 2 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 7 | 11 | 9 | 11 | 47
  White | 45 | 45 | 41 | 44 | 42 | 217
  More than one race | 1 | 1 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Hemagglutination Inhibition (HI) Antibody Response to the Vaccine Strain (A/H9N2/Chicken/Hong Kong/G9/97) Associated With Seroconversion 21 Days After the Second Vaccination
Time Frame: 21 days after 2nd vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg | 7.5 µg | 15 µg | 30 µg | 45 µg
Number analyzed (Participants) | 52 | 53 | 52 | 53 | 54
Participants | 27 | 27 | 38 | 41 | 48

2. Primary Outcome: Number of Subjects Achieving an HI Antibody Titer >= 1:40 21 Days After the Second Vaccination
Time Frame: 21 days after 2nd vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg | 7.5 µg | 15 µg | 30 µg | 45 µg
Number analyzed (Participants) | 52 | 53 | 52 | 53 | 54
Participants | 28 | 28 | 39 | 42 | 48

3. Primary Outcome: Number of Subjects With Injection Site and Systemic Reactions Within 7 Days After the First and Second Vaccination (Vacc) by Severity
Time Frame: 7 days after 1st and 2nd vaccination
Population: Participant number differs from 1st to 2nd vaccination due to dropouts
Measure: Number; unit: participants
Arm/Group | 3.75 µg | 7.5 µg | 15 µg | 30 µg | 45 µg
Number analyzed (Participants) | 56 | 55 | 54 | 55 | 55
participants
  Number of subjects with injection site reactions within 7 days after 1st vaccination : Mild | 9 | 10 | 16 | 17 | 20
  Number of subjects with injection site reactions within 7 days after 1st vaccination : Moderate | 0 | 0 | 3 | 0 | 3
  Number of subjects with injection site reactions within 7 days after 1st vaccination : Severe | 0 | 0 | 0 | 0 | 0
  Number of subjects with injection site reactions within 7 days after 1st vaccination : Unknown | 0 | 0 | 0 | 1 | 0
  Number of subjects with injection site reactions within 7 days after 2nd vaccination : Mild: number analyzed (Participants) | 53 | 53 | 54 | 55 | 54
  Number of subjects with injection site reactions within 7 days after 2nd vaccination : Mild | 6 | 8 | 14 | 10 | 18
  Number of subjects with injection site reactions within 7 days after 2nd vaccination : Moderate: number analyzed (Participants) | 53 | 53 | 54 | 55 | 54
  Number of subjects with injection site reactions within 7 days after 2nd vaccination : Moderate | 1 | 0 | 0 | 2 | 2
  Number of subjects with injection site reactions within 7 days after 2nd vaccination : Severe: number analyzed (Participants) | 53 | 53 | 54 | 55 | 54
  Number of subjects with injection site reactions within 7 days after 2nd vaccination : Severe | 0 | 0 | 1 | 0 | 0
  Number of subjects with injection site reactions within 7 days after 2nd vaccination : Unknown: number analyzed (Participants) | 53 | 53 | 54 | 55 | 54
  Number of subjects with injection site reactions within 7 days after 2nd vaccination : Unknown | 0 | 0 | 0 | 0 | 0
  Number of subjects with systemic reactions within 7 days after 1st vaccination : Mild | 6 | 13 | 12 | 10 | 11
  Number of subjects with systemic reactions within 7 days after 1st vaccination: Moderate | 0 | 1 | 2 | 1 | 2
  Number of subjects with systemic reactions within 7 days after 1st vaccination : Severe | 1 | 0 | 0 | 0 | 0
  Number of subjects with systemic reactions within 7 days after 1st vaccination : Unknown | 0 | 0 | 0 | 0 | 0
  Number of subjects with systemic reactions within 7 days after 2nd vaccination : Mild: number analyzed (Participants) | 53 | 53 | 54 | 55 | 54
  Number of subjects with systemic reactions within 7 days after 2nd vaccination : Mild | 3 | 3 | 7 | 4 | 3
  Number of subjects with systemic reactions within 7 days after 2nd vaccination: Moderate: number analyzed (Participants) | 53 | 53 | 54 | 55 | 54
  Number of subjects with systemic reactions within 7 days after 2nd vaccination: Moderate | 1 | 2 | 0 | 1 | 0
  Number of subjects with systemic reactions within 7 days after 2nd vaccination : Severe: number analyzed (Participants) | 53 | 53 | 54 | 55 | 54
  Number of subjects with systemic reactions within 7 days after 2nd vaccination : Severe | 0 | 0 | 0 | 0 | 0
  Number of subjects with systemic reactions within 7 days after 2nd vaccination : Unknown: number analyzed (Participants) | 53 | 53 | 54 | 55 | 54
  Number of subjects with systemic reactions within 7 days after 2nd vaccination : Unknown | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Subjects Achieving an HI Antibody Titer >= 1:40 21 Days After the First Vaccination
Time Frame: 21 days after 1st vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg | 7.5 µg | 15 µg | 30 µg | 45 µg
Number analyzed (Participants) | 56 | 54 | 54 | 55 | 54
Participants | 17 | 22 | 33 | 35 | 40

5. Secondary Outcome: Number of Subjects With Antibody Response Associated With Protection 21 Days After the First and Second Vaccination Defined as Microneutralization (MN) Titer >= 1:20
Time Frame: 21 days after 1st and 2nd vaccination
Population: Participant number differs from 1st to 2nd vaccination due to dropouts
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg | 7.5 µg | 15 µg | 30 µg | 45 µg
Number analyzed (Participants) | 56 | 54 | 54 | 55 | 54
Participants
  21 days after 1st vaccination | 45 | 48 | 49 | 55 | 54
  21 days after 2nd vaccination: number analyzed (Participants) | 52 | 53 | 52 | 53 | 54
  21 days after 2nd vaccination | 51 | 51 | 50 | 53 | 54

6. Secondary Outcome: Number of Subjects With Antibody Response Associated With Protection 21 Days After the First and Second Vaccination Defined as Single Radial Hemolysis (SRH) Area >= 25 mm2
Time Frame: 21 days after 1st and 2nd vaccination
Population: Participant number differs from 1st to 2nd vaccination due to dropouts
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg | 7.5 µg | 15 µg | 30 µg | 45 µg
Number analyzed (Participants) | 56 | 54 | 54 | 55 | 54
Participants
  21 days after 1st vaccination | 45 | 48 | 49 | 53 | 53
  21 days after 2nd vaccination: number analyzed (Participants) | 52 | 53 | 52 | 53 | 54
  21 days after 2nd vaccination | 49 | 52 | 51 | 52 | 54

7. Secondary Outcome: Number of Participants With Antibody Response 21 Days After the First and Second Vaccination Measured by HI, MN and SRH Assays
Time Frame: 21 days after 1st and 2nd vaccination
Population: Participant number differs from 1st to 2nd vaccination due to dropouts
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg | 7.5 µg | 15 µg | 30 µg | 45 µg
Number analyzed (Participants) | 56 | 54 | 54 | 55 | 54
Participants
  Antibody response 21 days after the 1st vaccination : Measured by HI assay | 16 | 21 | 32 | 35 | 40
  Antibody response 21 days after the 1st vaccination : Measured by MN assay | 40 | 44 | 47 | 52 | 53
  Antibody response 21 days after the 1st vaccination : Measured by SRH area | 30 | 39 | 35 | 42 | 42
  Antibody response 21 days after the 2nd vaccination : Measured by HI assay: number analyzed (Participants) | 52 | 53 | 52 | 53 | 54
  Antibody response 21 days after the 2nd vaccination : Measured by HI assay | 27 | 27 | 38 | 41 | 48
  Antibody response 21 days after the 2nd vaccination : Measured by MN assay: number analyzed (Participants) | 52 | 53 | 52 | 53 | 54
  Antibody response 21 days after the 2nd vaccination : Measured by MN assay | 49 | 49 | 49 | 51 | 53
  Antibody response 21 days after the 2nd vaccination : Measured by SRH area: number analyzed (Participants) | 52 | 53 | 52 | 53 | 54
  Antibody response 21 days after the 2nd vaccination : Measured by SRH area | 35 | 42 | 38 | 43 | 44

8. Secondary Outcome: Fold Increase of Antibody Response 21 Days After the First and Second Vaccination as Compared to Baseline Measured by HI, MN and SRH Assays
Time Frame: 21 days after 1st and 2nd vaccination
Population: Participant number differs from 1st to 2nd vaccination due to dropouts
Measure: Geometric Mean (90% Confidence Interval); unit: Fold Change in Antibody Response
Arm/Group | 3.75 µg | 7.5 µg | 15 µg | 30 µg | 45 µg
Number analyzed (Participants) | 56 | 54 | 54 | 55 | 54
Fold Change in Antibody Response
  Fold increase of antibody response measured after 1st vaccination by HI assay | 3.2 [2.5 to 4.1] | 4.5 [3.3 to 6.2] | 7.8 [5.8 to 10.5] | 10.4 [7.4 to 14.6] | 15.5 [11.7 to 20.5]
  Fold increase of antibody response measured after 2nd vaccination by HI assay: number analyzed (Participants) | 52 | 53 | 52 | 53 | 54
  Fold increase of antibody response measured after 2nd vaccination by HI assay | 5.7 [4.5 to 7.2] | 6.6 [5.0 to 8.7] | 10.7 [8.0 to 14.2] | 12.7 [9.7 to 16.8] | 19.8 [15.5 to 25.3]
  Fold increase of antibody response measured after 1st vaccination by MN assay | 8 [5.9 to 10.8] | 14.4 [10.3 to 20.3] | 18.9 [13.4 to 26.7] | 26.7 [19.3 to 36.8] | 44.1 [32.4 to 60.1]
  Fold increase of antibody response measured after 2nd vaccination by MN assay: number analyzed (Participants) | 52 | 53 | 52 | 53 | 54
  Fold increase of antibody response measured after 2nd vaccination by MN assay | 22.2 [17.2 to 28.6] | 25.5 [18.5 to 34.9] | 34.0 [25.2 to 45.9] | 38.9 [28.9 to 52.5] | 67.4 [51.1 to 88.8]
  Fold increase of antibody response measured after 1st vaccination by SRH assay | 2.7 [2.2 to 3.3] | 3.9 [3.0 to 4.9] | 3.2 [2.5 to 4.0] | 4.0 [3.2 to 5.1] | 5.1 [4.0 to 6.6]
  Fold increase of antibody response measured after 2nd vaccination by SRH assay: number analyzed (Participants) | 52 | 53 | 52 | 53 | 54
  Fold increase of antibody response measured after 2nd vaccination by SRH assay | 3.7 [2.9 to 4.6] | 4.5 [3.5 to 5.8] | 3.7 [2.9 to 4.7] | 4.4 [3.5 to 5.6] | 5.5 [4.3 to 7.2]

9. Secondary Outcome: Number of Subjects With Seroconversion (as Defined for the Primary Immunogenicity Endpoint) Measured by HI Assay 21 Days After the First Vaccination as Compared to Baseline
Time Frame: 21 days after 1st vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg | 7.5 µg | 15 µg | 30 µg | 45 µg
Number analyzed (Participants) | 56 | 54 | 54 | 55 | 54
Participants | 16 | 21 | 32 | 35 | 40

10. Secondary Outcome: Number of Subjects With Seroconversion Defined as a Minimum Fourfold Increase in Titer Measured by MN Assay 21 Days After the First and Second Vaccination as Compared to Baseline
Time Frame: 21 days after 1st and 2nd vaccination
Population: Participant number differs from 1st to 2nd vaccination due to dropouts
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg | 7.5 µg | 15 µg | 30 µg | 45 µg
Number analyzed (Participants) | 56 | 54 | 54 | 55 | 54
Participants
  Number of subjects with seroconversion 21 days after 1st vaccination | 40 | 44 | 47 | 52 | 53
  Number of subjects with seroconversion 21 days after 2nd vaccination: number analyzed (Participants) | 52 | 53 | 52 | 53 | 54
  Number of subjects with seroconversion 21 days after 2nd vaccination | 49 | 49 | 49 | 51 | 53

11. Secondary Outcome: Number of Subjects With Seroconversion as Measured by SRH Assay 21 Days After the First and Second Vaccination
Time Frame: 21 days after 1st and 2nd vaccination
Population: Participant number differs from 1st to 2nd vaccination due to dropouts
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg | 7.5 µg | 15 µg | 30 µg | 45 µg
Number analyzed (Participants) | 56 | 54 | 54 | 55 | 54
Participants
  Number of subjects with seroconversion 21 days after the 1st vaccination | 30 | 39 | 35 | 42 | 42
  Number of subjects with seroconversion 21 days after the 2nd vaccination: number analyzed (Participants) | 52 | 53 | 52 | 53 | 54
  Number of subjects with seroconversion 21 days after the 2nd vaccination | 35 | 42 | 38 | 43 | 44

12. Secondary Outcome: Number of Subjects With Antibody Response Associated With Protection 180 Days After the First Vaccination as Measured by HI, MN and SRH Assays
Time Frame: 180 days after 1st vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg | 7.5 µg | 15 µg | 30 µg | 45 µg
Number analyzed (Participants) | 51 | 51 | 51 | 51 | 52
Participants
  Subjects with antibody response 180 days after the 1st vaccination as measured by HI Assay | 10 | 17 | 22 | 28 | 31
  Subjects with antibody response 180 days after the 1st vaccination as measured by MN Assay | 38 | 43 | 45 | 49 | 52
  Subjects with antibody response 180 days after the 1st vaccination as measured by SRH Assay | 46 | 49 | 50 | 51 | 51

13. Secondary Outcome: Number of Subjects With Antibody Response 180 Days After the First Vaccination Measured by HI, MN and SRH Assays
Time Frame: 180 days after 1st vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | 3.75 µg | 7.5 µg | 15 µg | 30 µg | 45 µg
Number analyzed (Participants) | 51 | 51 | 51 | 51 | 52
Participants
  Subjects with antibody response 180 days after the 1st vaccination as measured by HI Assay | 9 | 17 | 21 | 28 | 31
  Subjects with antibody response 180 days after the 1st vaccination as measured by MN Assay | 34 | 41 | 44 | 47 | 52
  Subjects with antibody response 180 days after the 1st vaccination as measured by SRH Assay | 30 | 43 | 36 | 43 | 40

14. Secondary Outcome: Fold Increase of Antibody Response 180 Days After the First Vaccination as Compared to Baseline Measured by HI, MN and SRH Assays
Time Frame: 180 days after 1st vaccination
Measure: Geometric Mean (90% Confidence Interval); unit: Fold change in Antibody Response
Arm/Group | 3.75 µg | 7.5 µg | 15 µg | 30 µg | 45 µg
Number analyzed (Participants) | 51 | 51 | 51 | 51 | 52
Fold change in Antibody Response
  Fold increase of antibody response measured by HI Assay | 2.7 [2.2 to 3.2] | 3.9 [3.0 to 5.1] | 4.3 [3.4 to 4.6] | 6.1 [4.9 to 7.6] | 8.1 [6.6 to 9.9]
  Fold increase of antibody response measured by MN Assay | 5.4 [4.2 to 7.0] | 9.1 [6.5 to 12.7] | 10.3 [7.9 to 13.3] | 13.3 [10.3 to 17.2] | 19.9 [15.4 to 25.8]
  Fold increase of antibody response measured by SRH Assay | 3.4 [2.7 to 4.3] | 4.5 [3.5 to 5.8] | 3.7 [2.9 to 4.7] | 4.5 [3.5 to 5.7] | 5.1 [4.0 to 6.6]

15. Secondary Outcome: Number of Subjects With Fever, Malaise and Shivering With Onset Within 7 Days After the First and Second Vaccination
Time Frame: 7 days after 1st and 2nd vaccination
Population: Participant number differs from 1st to 2nd vaccination due to dropouts
Measure: Count of Participants; unit: Participants
Groups:
- 40 µg: Subjects to receive 2 intramuscular injections of Reverse Genetic (RG) reassortant A/H9N2 influenza vaccine on Day 1 and Day 22
Arm/Group | 3.75 µg | 7.5 µg | 15 µg | 30 µg | 40 µg
Number analyzed (Participants) | 56 | 55 | 54 | 55 | 55
Participants
  After 1st vaccination : Fever | 0 | 0 | 0 | 0 | 0
  After 1st vaccination : Malasie | 1 | 2 | 2 | 1 | 2
  After 1st vaccination : Shivering | 0 | 3 | 0 | 0 | 2
  After 2nd vaccination : Fever: number analyzed (Participants) | 53 | 53 | 54 | 55 | 54
  After 2nd vaccination : Fever | 0 | 0 | 0 | 0 | 1
  After 2nd vaccination : Malasie: number analyzed (Participants) | 53 | 53 | 54 | 55 | 54
  After 2nd vaccination : Malasie | 0 | 2 | 3 | 0 | 0
  After 2nd vaccination : Shivering: number analyzed (Participants) | 53 | 53 | 54 | 55 | 54
  After 2nd vaccination : Shivering | 1 | 0 | 0 | 0 | 0

16. Secondary Outcome: Frequency and Severity of Adverse Events (AEs) Observed During the Entire Study Period
Time Frame: Through study completion by all subjects, an average of 181 days (+/- 14 days)
Measure: Number; unit: Events
Arm/Group | 3.75 µg | 7.5 µg | 15 µg | 30 µg | 45 µg
Number analyzed (Participants) | 56 | 55 | 54 | 55 | 55
Events
  Mild | 25 | 54 | 67 | 46 | 64
  Moderate | 2 | 5 | 7 | 4 | 10
  Severe | 2 | 0 | 1 | 0 | 0
  Unknown | 0 | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Arm/Group | 3.75 µg | 7.5 µg | 15 µg | 30 µg | 45 µg
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/55 | 0/54 | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/55 | 0/54 | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 15/56 | 23/55 | 27/54 | 27/55 | 28/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 3.75 µg (N=56) | 7.5 µg (N=55) | 15 µg (N=54) | 30 µg (N=55) | 45 µg (N=55)
Injection Site Reactions (General disorders) | 9 | 11 | 20 | 18 | 26 — After 1st vaccination
Injection Site Reactions (General disorders) | 7/53 | 8/53 | 15 | 12 | 20/54 — After 2nd vaccination
Fatigue (General disorders) | 3 | 9 | 4 | 2 | 2 — After 1st vaccination
Malaise (General disorders) | 1 | 2 | 2 | 1 | 2 — After 1st vaccination
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 — After 1st vaccination
Aspartate aminotransferase (Investigations) | 1 | 0 | 1 | 1 | 0 — After 1st vaccination
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 3 | 5 — After 1st vaccination
Headache (Nervous system disorders) | 2 | 9 | 10 | 4 | 6 — After 1st vaccination
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 — After 1st vaccination
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 — After 1st vaccination
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 — After 1st vaccination
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 — After 1st vaccination
Chills (General disorders) | 0 | 2 | 0 | 0 | 2 — After 1st vaccination
Hyperhidrosis (General disorders) | 0 | 1 | 0 | 0 | 1 — After 1st vaccination
General pain (General disorders) | 0 | 1 | 0 | 0 | 0 — After 1st vaccination
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 — After 1st vaccination
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 — After 1st vaccination
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 1 | 1 — After 1st vaccination
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 — After 1st vaccination
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 — After 1st vaccination
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 — After 1st vaccination
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 — After 1st vaccination
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 1 — After 1st vaccination
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 — After 1st vaccination
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 — After 1st vaccination
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 — After 1st vaccination
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 — After 1st vaccination
Fatigue (Eye disorders) | 1/53 | 3/53 | 3 | 1 | 2/54 — After 2nd vaccination
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/53 | 0/53 | 1 | 0 | 0/54 — After 2nd vaccination
Myalgia (Musculoskeletal and connective tissue disorders) | 1/53 | 1/53 | 3 | 0 | 1/54 — After 2nd vaccination
Headache (Nervous system disorders) | 3/53 | 1/53 | 2 | 4 | 1/54 — After 2nd vaccination
Malaise (General disorders) | 0/53 | 2/53 | 3 | 0 | 0/54 — After 2nd vaccination
Nausea (Gastrointestinal disorders) | 0/53 | 0/53 | 1 | 0 | 0/54 — After 2nd vaccination
Hyperhidrosis (General disorders) | 0/53 | 0/53 | 2 | 0 | 0/54 — After 2nd vaccination
Irritability (General disorders) | 0/53 | 0/53 | 1 | 0 | 0/54 — After 2nd vaccination
Dizziness (Nervous system disorders) | 0/53 | 0/53 | 2 | 0 | 0/54 — After 2nd vaccination
Dysgeusia (Nervous system disorders) | 0/53 | 0/53 | 1 | 0 | 0/54 — After 2nd vaccination
Rash generalised (Skin and subcutaneous tissue disorders) | 0/53 | 0/53 | 0 | 1 | 0/54 — After 2nd vaccination
Body temp increased (Investigations) | 0 | 0 | 1 | 0 | 0 — After 2nd vaccination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No